CLINICAL TRIAL: NCT04616391
Title: Transition of Patients With T1D From Multiple Daily Injection (MDI) and Self-Monitoring of Blood Glucose (SMBG) Directly to MiniMed™ 780G Advanced Hybrid Closed Loop (AHCL) System :Impact on Glucose Control and Quality of Life Measures
Brief Title: AHCL System Initiation in T1D Patients naïve to Technology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jagiellonian University (Other)
Collaborators: Medtronic Poland Spółka z ograniczoną odpowiedzialnością (Industry); University of Rzeszow (Other)
Responsible Party: Principal Investigator, Tomasz Klupa, Prof, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1072.61201.8.2020
Record Dates: First submitted 2020-10-29; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Medtronic 780G; Continous glucose monitoring systems; Insulin pump; diabetes type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: The trial is a two-centers, randomized controlled, parallel group study. Patients will be followed up during approximatively 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MDI group: (No Intervention): The patient continues MDI treatment as per routine procedures
- AHCL group (Experimental): The patient will use MiniMed 780G AHCL system
  Interventions: Device: insulin pump Medtronic 780G

INTERVENTIONS:
Device: insulin pump Medtronic 780G — Patients from the AHCL group will use the MiniMed 780G AHCL system. This system is already CE-marked.
  The AHCL system will be initiated first in Manual Mode (i.e. without AHCL control) with suspend before low feature (Visit 1).
  The AHCL system will be initiated in Auto Mode (i.e. with AHCL control) at Visit 2 with the settings in the below table. The Insulin to Carb ratio (ICR) and the Active Insulin Time (AIT) may be adjusted by the physician during the study. The glucose target may not be adjusted, unless in case of safety concerns. The patients may not adjust system settings without consulting with the physician.
  At each visit, the AHCL system data will be downloaded and reviewed by the physician. The patient interaction with the system will be evaluated, included sensor calibration, bolus management (before the meals and for corrections as needed), alarms and Auto Mode exits.
  Arms: AHCL group

SUMMARY:
The primary objective of this study is to evaluate whether the MiniMed 780G AHCL system improves glycemic control and Quality of Life (QoL) perception in adult individuals with T1D and naïve to CSII and CGM technologies.

The trial is a two-centers, randomized controlled, parallel group study. Patients will be followed up during approximatively 3 months.

DETAILED DESCRIPTION:
Recent advances in insulin pumps, continuous glucose monitoring (CGM) devices, and control algorithms have resulted in an acceleration of progress in the development of the automated systems of insulin delivery including hybrid closed loop (HCL) systems.

Initial studies on the MiniMed 670G system, the first HCL system approved, have reported increased glycemic control in both adults and pediatrics, having experience with insulin pump therapy with or without experience of CGM technology. More recently it was shown shown even further improvement in glycemic control with the 670G system, in children and adolescents naïve to both pump and CGM technologies. This may be, at least partially, due to lack of willingness of patients to "let the algorithm work" based on their previous experience with CSII and CGM.

The investigators aim to evaluate the impact of an Advanced Hybrid Closed Loop (AHCL) system in adults naïve to pump and CGM technology. For this purpose the investigators target the population of T1DM individuals who are older than 26 years. The study will be conducted in Poland, where only individuals under the age of 26 are entitled to CSII/CGM reimbursement.

If the study succeeds in terms of improved glycemic patterns, quality of life and patients' acceptance, it may provide evidence for consideration in CSII/CGM reimbursement for this population.

Devices usage in the study:

Envision Pro device (CE-marked) will be used to collect CGM data in a retrospective manner. Envision Pro records up to 6 days of data. Patients will wear 2 consecutive Envision Pro devices both during the run-in phase and the at the end of the study phase, i.e. up to 12 days of data. The first Envision Pro device will be placed in the hospital and the second Envision Pro device will be placed by the patient at home, assisted by the study staff on the phone.

In addition, patients from the AHCL group will use the MiniMed 780G AHCL system (CE-marked). The AHCL system will be initiated first in Manual Mode (i.e. without AHCL control) with suspend before low feature. In short, the protocol inputs the current insulin program (MDI) and calculates a 10-20% reduction in total daily dose, with a 40/60 basal/bolus distribution in four or five basal rates. Insulin-to-carbohydrate ratio (ICR) settings utilize the formula of 300-450/total daily dose (TDD) and the formula of 90-110/TDD (mmol/L) with two CF settings; the nighttime CF factor is set 10-20% higher than the daytime CF. Active insulin is set time (3 h); suspend before low feature is turned on with a threshold of 3.0-3.8 mmol/L (55-70 mg/dL), and glucose target ranges from 5.0 to 7.2 mmol/L (90-130 mg/dL.

The AHCL system will be initiated in Auto Mode (i.e. with AHCL control) at Visit 2.At each visit, the AHCL system data will be downloaded and reviewed by the physician. The patient interaction with the system will be evaluated, included sensor calibration, bolus management (before the meals and for corrections as needed), alarms and Auto Mode exits.

At each visit, the glycemic control will be reviewed, and system settings re-assessed and adjusted as needed, including ICR, AIT and basal rates in Manual Mode.

The trial is a two-centers, randomized controlled, parallel group study. Patients will be followed up during approximatively 3 months.

Study phase

Both groups will have a similar number of visits in order to minimize bias. However, the AHCL group will have 2 additional visits to allow for patients to be trained on the AHCL system.

MDI group:

The patient continues MDI treatment as per routine procedures

* Visit 1 (day 0, can be combined with the randomization visit): BG meter data download, data review and optimization of MDI management.
* Visit 2 (Visit 1 + 14 days, window +/- 3 days): BG meter data download, data review and optimization of MDI management
* Visit 3 (Visit 2 + 14 days, window +/- 3 days): BG meter data download, data review and optimization of MDI management
* Visit 4 (Visit 3 + 28 days, window +/- 7 days): BG meter data download, data review and optimization of MDI management
* Visit 5 Visit 4 + 22 days, window +/- 7 days): BG meter data download, data review and optimization of MDI management, first professional CGM evaluation start.
* Visit 6 (Visit 5 + 6 days, window +3 days) - phone call: second professional CGM evaluation start.
* Visit 7 (Visit 9 + 6 days, window + 3 days): QoL questionnaire, blood sample for HbA1c lab test.

Professional CGM evaluation will be repeated for 6 days in cased less than 10 days data is available.

Study conclusion.

AHCL group:

* Visit 1 (day 0, can be combined with the randomization visit): the patient will get the pre-reading materials on the 780G system, to be read before Visit 2. CGM training and initiation.
* Visit 2 (Visit 1 + 1 day, window +7 days): 780G system training and initiation in Manual Mode.
* Visit 3 (Visit 2 +3 days, window +3 days): 780G system data download. Auto Mode readiness assessment. 780G system initiation in Auto Mode with AHCL control
* Visit 4 (Visit 3 + 3 days, window +1 day) - phone call: Auto Mode initiation follow-up.
* Visit 5 (Visit 4 + 7 days, window +/- 3 days): 780G system data download, therapy assessment and optimization
* Visit 6 (Visit 5 + 14 days, window +/- 3 days): 780G system data download, therapy assessment and optimization
* Visit 7 (Visit 6 + 28 days, window +/- 7 days): 780G system data download, therapy assessment and optimization
* Visit 8 (Visit 7 + 22 days, window +/- 7 days): 780G system data download, therapy assessment and optimization, first professional CGM evaluation start.
* Visit 9 (Visit 8 + 6 days, window +3 days) - phone call: second professional CGM evaluation start.
* Visit 10 (Visit 9 + 6 days, window + 3 days): 780G system data download, QoL questionnaire, blood sample for HbA1c lab test.

Professional CGM evaluation will be repeated for 6 days in cased less than 10 days data is available.

Study Conclusion

Study endpoints

* Between group comparison of data measured by CGM technology will be performed based on data collected by professional CGM in both groups.
* Between group comparison of Quality of Life.

ELIGIBILITY:
Inclusion Criteria:

1. Age 26 - 60 years at time of screening a clinical diagnosis of type 1 diabetes for 2 years or more as determined via medical record or source documentation by an individual qualified to make a medical diagnosis
2. Willing to participate in a study for the specified duration
3. Willing to perform ≥ 4 finger stick blood glucose measurements daily
4. Willing to perform required sensor calibrations
5. Willing to wear the system continuously throughout the study
6. Glycosylated hemoglobin (A1C) value less than 10.0% at time of screening visit
7. Treated with MDI
8. Willing to perform at least 4 BGM/day, when on MDI
9. At least communicative level of English to be able to understand the pump interface.

Exclusion Criteria:

1. Previous treatment with CSII/CGM
2. Usage of ultra-rapid insulins, e.g. FIASP
3. concurrent illness
4. laboratory abnormalities, or medications that might affect study participation,
5. current pregnancy
6. renal impairment
7. hemoglobin A1c value above 10%.

Ages: 26 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-11-02 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Between group TIR difference | Day 78-90
  Between group difference in the percentage of time spent within range with sensor glucose (SG) between 70-180 mg/dL (TIR) (3.9-10.0 mmol/L).

SECONDARY OUTCOMES:
Between group TIR difference >70% | Day 78-90
  Between groups difference in the percentage of participants achieving TIR >70%
Between group difference in the percentage of time spent: | Day 78-90
  • Between group difference in the percentage of time spent:
  * in hyperglycemic range with SG > 250 mg/dL (13.9 mmol/L)
  * in hyperglycemic range with SG > 180 mg/dL (10.0 mmol/L)
  * in hypoglycemic range with SG < 54 mg/dL (3.0 mmol/L)
  * in hypoglycemic range with SG < 70 mg/dL (3.9 mmol/L)
Between group difference in the mean glucose level | Day 78-90
  Between group difference in the mean glucose level
Between group difference in the glycemic variability measure by SD and CV | Day 78-90
  Between group difference in the glycemic variability measure by SD and CV
Between group difference in the HbA1c levels | Day 78-90
  Between group difference in the HbA1c levels
Between group difference in the Diabetes Quality of Life (QoL) questionnaire score | Day 90
  Between group difference in the Diabetes Quality of Life (QoL) questionnaire score

OTHER OUTCOMES:
Number of severe hypoglycemic episodes | Day 90
  "Severe Hypoglycemia" is an event requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. These episodes may be associated with sufficient neuroglycopenia to induce seizure or coma. Plasma glucose measurements may not be available during such an event, but neurological recovery attributable to the restoration of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration. (American Diabetes Association Workgroup on Hypoglycemia, Diabetes Care 28:1245-1249, 2005)
Number of Diabetic Ketoacidosis events | Day 90
  "Diabetic Ketoacidosis/DKA" is defined as: Hyperglycemia (blood glucose >250 mg/dL or >13.9 mmol/L) with either low serum bicarbonate (<15 mEq/L) and/or low pH (<7.24) Anion gap (> 12) and either ketonemia or ketonuria and requiring treatment within a health-care facility. (American Diabetes Association-Diabetes Care, Volume 27, Supplement 1, January 2004).
Number of Severe Hyperglycemia episodes | Day 90
  "Severe Hyperglycemia" is defined as Hyperglycemia (blood glucose >270 mg/dL) with blood glucose ketones >0.6mmol/L or accompanied by symptoms of nausea, vomiting or abdominal pain.

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Klupa, Prof, Principal Investigator — Hospital University; jagiellonian University Medical College

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bergenstal RM, Garg S, Weinzimer SA, Buckingham BA, Bode BW, Tamborlane WV, Kaufman FR. Safety of a Hybrid Closed-Loop Insulin Delivery System in Patients With Type 1 Diabetes. JAMA. 2016 Oct 4;316(13):1407-1408. doi: 10.1001/jama.2016.11708. No abstract available. PMID 27629148
- [Result] Cordero TL, Garg SK, Brazg R, Bailey TS, Shin J, Lee SW, Kaufman FR. The Effect of Prior Continuous Glucose Monitoring Use on Glycemic Outcomes in the Pivotal Trial of the MiniMed 670G Hybrid Closed-Loop System. Diabetes Technol Ther. 2017 Dec;19(12):749-752. doi: 10.1089/dia.2017.0208. Epub 2017 Nov 17. PMID 29148821
- [Result] Forlenza GP, Messer LH, Berget C, Wadwa RP, Driscoll KA. Biopsychosocial Factors Associated With Satisfaction and Sustained Use of Artificial Pancreas Technology and Its Components: a Call to the Technology Field. Curr Diab Rep. 2018 Sep 26;18(11):114. doi: 10.1007/s11892-018-1078-1. PMID 30259309
- [Result] Petrovski G, Al Khalaf F, Campbell J, Fisher H, Umer F, Hussain K. 10-Day structured initiation protocol from multiple daily injection to hybrid closed-loop system in children and adolescents with type 1 diabetes. Acta Diabetol. 2020 Jun;57(6):681-687. doi: 10.1007/s00592-019-01472-w. Epub 2020 Jan 17. PMID 31953687
- [Result] Beck RW, Riddlesworth T, Ruedy K, Ahmann A, Bergenstal R, Haller S, Kollman C, Kruger D, McGill JB, Polonsky W, Toschi E, Wolpert H, Price D; DIAMOND Study Group. Effect of Continuous Glucose Monitoring on Glycemic Control in Adults With Type 1 Diabetes Using Insulin Injections: The DIAMOND Randomized Clinical Trial. JAMA. 2017 Jan 24;317(4):371-378. doi: 10.1001/jama.2016.19975. PMID 28118453
- [Derived] Cyranka K, Matejko B, Juza A, Kiec-Wilk B, Krzyzowska S, Cohen O, Da Silva J, Lushchyk M, Malecki MT, Klupa T. Improvement of Selected Psychological Parameters and Quality of Life of Patients With Type 1 Diabetes Mellitus Undergoing Transition From Multiple Daily Injections and Self-Monitoring of Blood Glucose Directly to the MiniMed 780G Advanced Hybrid Closed-Loop System: Post hoc Analysis of a Randomized Control Study. JMIR Form Res. 2023 Jan 24;7:e43535. doi: 10.2196/43535. PMID 36692945
- [Derived] Cyranka K, Matejko B, Chrobak A, Dudek D, Kiec-Wilk B, Cyganek K, Witek P, Lushchyk M, Krzyzowska S, Malecki MT, Klupa T. Assessment of the spectrum of depression and bipolarity in patients with type 1 diabetes. Diabetes Metab Res Rev. 2023 Jan;39(1):e3583. doi: 10.1002/dmrr.3583. Epub 2022 Nov 6. PMID 36270020